CLINICAL TRIAL: NCT07360262
Title: Time-dependent Recovery of Gastric Emptying After Cessation of Glucagon-like Peptide-1 Receptor Agonists: a Prospective Observational Gastric Ultrasound Study
Brief Title: Gastric Emptying Recovery After GLP-1 RA Cessation
Status: Completed | Type: Observational
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor, Wonkwang University Hospital
Other Study IDs: Wonkwang UH 23
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Gastric Emptying; Gastroparesis; Preoperative Care
Keywords: GLP-1 receptor agonist; GLP-1 RA cessation / withholding interval; Point-of-care ultrasound / POCUS; Gastric ultrasound; Residual gastric volume
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GLP-1 RA cessation ≤3 days: Participants using GLP-1 receptor agonists whose last dose was taken ≤3 days before the preoperative gastric ultrasound assessment (performed immediately prior to induction of anesthesia).
  Interventions: Other: Preoperative gastric ultrasound
- GLP-1 RA cessation 4-7 days: Participants using GLP-1 receptor agonists whose last dose was taken 4-7 days before the preoperative gastric ultrasound assessment (performed immediately prior to induction of anesthesia).
  Interventions: Other: Preoperative gastric ultrasound
- GLP-1 RA cessation ≥8 days: Participants using GLP-1 receptor agonists whose last dose was taken ≥8 days before the preoperative gastric ultrasound assessment (performed immediately prior to induction of anesthesia).
  Interventions: Other: Preoperative gastric ultrasound

INTERVENTIONS:
Other: Preoperative gastric ultrasound — Preoperative point-of-care gastric ultrasound was performed immediately prior to induction of anesthesia to assess qualitative gastric content and to estimate gastric volume from antral cross-sectional area. The procedure was observational and was applied to all cohorts; no study-assigned treatment was administered or modified.
  Other Names: Point-of-care gastric ultrasound (Gastric POCUS)

SUMMARY:
Glucagon-like peptide-1 receptor agonists (GLP-1 RAs) can delay gastric emptying and may increase residual gastric contents before general anesthesia. Current perioperative recommendations for withholding GLP-1 RAs (e.g., a fixed 7-day discontinuation for weekly agents) are largely consensus-based, and it is unclear whether gastric emptying normalizes abruptly after a single threshold interval. This prospective observational cohort study will evaluate how preoperative residual gastric content changes with increasing time since the last GLP-1 RA dose, using point-of-care gastric ultrasound performed immediately before induction of anesthesia. Time since last dose will be analyzed as a continuous exposure and across prespecified intervals (≤3 days, 4-7 days, ≥8 days). The primary outcome is ultrasound-estimated gastric volume normalized to body weight (mL/kg), derived from antral cross-sectional area. Secondary outcomes include the presence of a "high-risk stomach" based on gastric volume criteria and qualitative ultrasound findings. The study will also assess whether body mass index modifies the relationship between cessation interval and gastric volume, thereby supporting individualized perioperative risk assessment.

DETAILED DESCRIPTION:
Study design and setting: This is a prospective observational cohort study conducted at a tertiary academic hospital to evaluate gastric emptying recovery after cessation of GLP-1 receptor agonists. Adult patients (≥18 years) receiving GLP-1 RAs and scheduled for elective surgery under general anesthesia will be enrolled consecutively to minimize selection bias. Prespecified exclusions include prior gastric or esophageal surgery, known gastroparesis, severe gastroesophageal reflux disease, emergency surgery, pregnancy, and inability to provide informed consent.

Exposure (no intervention assignment): The study does not assign or modify GLP-1 RA therapy. Time since the last GLP-1 RA dose will be recorded in days using patient report and medical records and analyzed both as a continuous variable and as prespecified categories (≤3 days, 4-7 days, ≥8 days). Information on GLP-1 RA formulation (weekly vs daily) and dose equivalence may be collected for sensitivity analyses. Potential confounders such as fasting duration and type of surgery will be recorded.

Gastric ultrasound procedures: Point-of-care gastric ultrasound will be performed immediately before induction of anesthesia using a standardized protocol by trained consultant anesthesiologists. The gastric antrum will be assessed in the supine and right lateral decubitus positions. Qualitative assessment of gastric content will be documented, and quantitative measurements of antral cross-sectional area will be used to estimate gastric volume.

Outcomes: The primary outcome is estimated gastric volume normalized to body weight (mL/kg). Secondary outcomes include the presence of a high-risk stomach, as defined by prespecified gastric volume criteria and qualitative ultrasound findings. Additional exploratory analyses will evaluate whether body mass index modifies the association between cessation interval and gastric volume and whether patient-reported gastrointestinal symptoms correlate with ultrasound findings.

Analysis overview: Associations between time since the last GLP-1 RA dose and gastric ultrasound outcomes will be assessed using prespecified regression models adjusted for relevant covariates (e.g., age, sex, BMI, diabetes status, fasting duration, and symptom measures). The interaction between BMI and cessation interval will be evaluated to characterize potential effect modification.

ELIGIBILITY:
Inclusion Criteria

* Adults aged ≥18 years
* Receiving a glucagon-like peptide-1 receptor agonist (GLP-1 RA)
* Scheduled for elective surgery under general anesthesia
* Able to provide written informed consent

Exclusion Criteria

* Prior gastric or esophageal surgery
* Known gastroparesis
* Severe gastroesophageal reflux disease
* Emergency surgery
* Pregnancy
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving GLP-1 receptor agonists who were scheduled for elective surgery under general anesthesia at a tertiary academic hospital and underwent preoperative point-of-care gastric ultrasound immediately prior to induction of anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2025-11-20 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
Ultrasound-estimated gastric volume (mL/kg) | Immediately preoperatively (just before induction of anesthesia)
  Estimated gastric volume normalized to body weight (mL/kg) was calculated from the gastric antral cross-sectional area measured by preoperative point-of-care ultrasound using validated equations.

SECONDARY OUTCOMES:
Perlas grade of gastric content (0-2) | Immediately preoperatively (just before induction of anesthesia)
  Qualitative gastric ultrasound grading of gastric content was recorded using the Perlas classification (Grade 0, 1, or 2) based on antral appearance in the supine and right lateral decubitus positions.
Antral cross-sectional area (CSA, cm²) | Immediately preoperatively (just before induction of anesthesia)
  Gastric antral cross-sectional area (cm²) was measured by preoperative ultrasound and used to estimate gastric volume.

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Lee, M.D.,Ph.D, Principal Investigator — Wonkwang University Hospital
Locations (2):
- South Korea (2):
  - Wonkwang University Hospital, Iksan, Jeollabuk-do
  - Wonkwang University School of Medicine Hospital, Iksan, Jeollabuk-do